CLINICAL TRIAL: NCT06358456
Title: Influence of Artificial Tears on Corneal Parameter Measurement Using Three Different Devices: Scheimpflug-, Keratometry - and Placido-technology
Brief Title: Influence of Artificial Tears on Keratometry and Biometry Measurements With Different Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Professor Dr. med. Thomas Kohnen, Prof. Dr. Thomas Kohnen, University Clinic Frankfurt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-928
Record Dates: First submitted 2024-03-12; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: artificial tears; keratometry; topography
MeSH Terms: interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: one arm for each diagnostic device (three in total)
Masking Description: The investigator and patient knew which device they were tested on
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IOL Master 700 (Active Comparator): Patients in this arm are measured twice with the IOL master 700 without intervention. After this artificial tears are applied and followed by 4 more measurements
  Interventions: Drug: Artificial tear; Other: No artificial tears
- Pentacam AXL (Active Comparator): Patients in this arm are measured twice with the Pentacam AXL without intervention. After this artificial tears are applied and followed by 4 more measurements
  Interventions: Drug: Artificial tear; Other: No artificial tears
- Galilei G6 (Active Comparator): Patients in this arm are measured twice with the Galilei G6 without intervention. After this artificial tears are applied and followed by 4 more measurements
  Interventions: Drug: Artificial tear; Other: No artificial tears

INTERVENTIONS:
Drug: Artificial tear — Application of low viscosity artificial tears (Artelac EDO). The active ingredient is hypromellose (1.92 mg per 0.6 ml container).
  Other Names: Artelac EDO
Other: No artificial tears — Before artificial tear application, 2 baseline measurements were taken of the cornea without any intervention

SUMMARY:
The goal of this clinical trial is to learn about the influence of artificial tears on measurements of healthy eyes with three different devices. The main questions it aims to answer are:

* Do artificial tears alter the measurements of the corneal surface
* Is there a difference between the devices used in this study

This is relevant because high quality measurements improve the postoperative outcome after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy eyes

Exclusion Criteria:

* Any prior intraocular surgery or trauma
* Any corneal pathology (ABMD, Fuch's, etc.)
* Active ocular pathology (e.g., amblyopia, ARMD)
* Contact lens wear within 2 weeks of study
* Any corneal relaxing incisions or astigmatic keratotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Does the application of artificial tears (Artelac EDO) alter the measurement of the anterior surface of the cornea (K mean in Diopters) using devices that either use keratometry or Scheimpflug-technology (IOL Master 700, Pentacam AXL or Galilei G6) | Comparison between the baseline measurements and the measurements 30 seconds after artificial tear application
  Difference of measurement of the mean corneal refractive power in diopters before artificial tear application and after artificial tear application using one of three devices (IOL Master 700, Pentacam AXL or Galilei G6)

SECONDARY OUTCOMES:
Is there any difference in anterior corneal refractive power measurements (K mean in Diopters) between the three different devices (IOL Master 700, Pentacam AXL, Galilei G6) after artificial tear (Artelac EDO) application? | Comparison between the baseline measurements and the measurements 30 seconds after artificial tear application
  Difference of measurement of the mean corneal refractive power in diopters before artificial tear (Artelac EDO) application and after artificial tear application between the three devices (IOL Master 700 using Keratometry, Pentacam AXL and Galilei G6 using Schmeipflug technology)
Does the application of artificial tears (Artelac EDO) alter the anterior astigmatism measurements (in diopters) using devices that either use keratometry or Scheimpflug-technology (IOL Master 700, Pentacam AXL or Galilei G6) | Comparison between the baseline measurements and the measurements 30 seconds after artificial tear application
  Difference of measurement of the mean corneal astigmatism in diopters before artificial tear (Artelac EDO) application and after artificial tear application using three different devices (IOL Master 700, Pentacam AXL and Galilei G6)
If there is an influence of artificial tears (Artelac EDO) on the measurement of the anterior surface of the cornea (K mean in Diopters) using the devices (IOL Master 700, Pentacam AXL or Galilei G6), how long does it last (in minutes)? | Comparison between the baseline measurements and the measurements up to 10 minutes after artificial tear applications
  How long does the difference of mean corneal refractive power in diopters before artificial tear (artelac ego) application and after artificial tear application last

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roggla V, Leydolt C, Schartmuller D, Schwarzenbacher L, Meyer E, Abela-Formanek C, Menapace R. Influence of Artificial Tears on Keratometric Measurements in Cataract Patients. Am J Ophthalmol. 2021 Jan;221:1-8. doi: 10.1016/j.ajo.2020.08.024. Epub 2020 Aug 21. PMID 32828877